CLINICAL TRIAL: NCT03988933
Title: 2R2: Higher Dose Rifampin for 2 Months vs Standard Dose Rifampin for Latent TB: a 3-arm Randomized Trial.
Brief Title: 2R2: Higher Dose Rifampin for 2 Months vs Standard Dose Rifampin for Latent TB.
Acronym: 2R2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dick Menzies, Senior Investigator at Research Institute of McGill University Health Center, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FND-143350-1
Record Dates: First submitted 2019-06-13; First posted 2019-06-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Latent Tuberculosis
Keywords: Latent Tuberculosis; Rifampin; Short Treatment for Latent Tuberculosis; High dose rifampin
MeSH Terms: conditions — Latent Tuberculosis | interventions — Rifampin

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1:1 to be in control arm or in one of the two intervention arms.
  Intervention arms:
  Arm 1: 60 doses daily self-administered rifampin at 20 mg/kg (2R20 - maximum 1200 mg/day).
  Arm 2: 60 doses daily self-administered rifampin at 30 mg/Kg (2R30) - maximum 1800 mg/day).
  Comparator:
  Arm 3 (standard): 120 doses daily self-administered rifampin at 10mg/kg (4R10maximum 600mg per day).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a partially double-blinded trial. Participation in control arm will be open label while participation in the two intervention arms will be double-blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Intervention Arm 1 (Experimental): Two months of daily self-administered rifampin at 20 mg/kg (maximum 1200 mg/day).
  Interventions: Drug: Rifampin double dose
- Intervention Arm 2 (Experimental): Two months of daily self-administered rifampin at 30 mg/Kg (maximum 1800 mg/day).
  Interventions: Drug: Rifampin triple dose
- Control Arm (Active Comparator): Four months of daily self-administered rifampin at a dose of 10mg per kg per day (maximum 600mg per day).
  Interventions: Drug: Rifampin standard dose

INTERVENTIONS:
Drug: Rifampin double dose — Double dose of rifampin for 2 months.
  Other Names: 2R20
  Arms: Intervention Arm 1
Drug: Rifampin triple dose — Triple dose of rifampin for 2 months.
  Other Names: 2R30
  Arms: Intervention Arm 2
Drug: Rifampin standard dose — Standard dose of rifampin for 4 months.
  Other Names: 4R10
  Arms: Control Arm

SUMMARY:
Rationale:

Shorter regimens of high dose daily rifampin may be safe, and as effective as the standard rifampin regimen when taken for 4 months to treat latent TB (LTBI). However, there is insufficient evidence on the optimal dose of rifampin that has similar efficacy as the standard 4-month rifampin regimen without jeopardizing safety or affecting completion rates.

Objectives:

The general purpose of this study is to determine if rifampin at double or triple the standard dose for 2 months is as safe and effective as the standard dose of rifampin when taken for 4 months to treat latent tuberculosis (TB).

Treatment:

Persons who need treatment for latent TB, will be given rifampin, either at the standard dose (10mg/kg/day) for 4 months (control arm); or at double dose (20mg/kg/day) for 2 months (intervention arm 1); or at triple dose (30mg/kg/day) for 2 months (intervention arm 2).

Design:

This is 1:1:1 randomized, phase 2b, partially blind, controlled trial. The two higher doses (intervention arms) will be administered double-blind: participants and providers will be aware of the duration of their regimen, but they will both remain blinded to the specific dose (i.e. 20 or 30 mg/kg/day) for those randomized to 2-months regimens. All members of the same household of a patient with newly diagnosed active pulmonary TB will be randomized together (i.e. cluster randomized).

Population and setting:

Adults and children aged 10 years and above, who have latent TB infection and are recommended by their doctor to take treatment for latent TB can participate in the study.

The planned number of persons with latent TB to recruit is about 1359 in total (or about 453 for each of the three arms).

The study will take place in 6 sites: four in Canada (Calgary, Edmonton, Montreal and Vancouver), one in Indonesia (Bandung) and one in Viet Nam (1 clinic in Ho Chi Min City and 3 clinics in Ha Noi).

Outcomes:

Primary outcomes are: 1) Treatment completion and 2) Safety (i.e. grade 3-5 adverse events).

Secondary outcomes are: 1) Safety (i.e. grade 1-2 adverse events) and 2) Efficacy (i.e. rates of active TB in the 26 months post-randomization). More information on how outcomes are defined is provided in the detailed description below.

DETAILED DESCRIPTION:
Additional information extracted from study protocol is provided below:

Study duration:

The study started in September 2019. Enrollment has started in all study sites and is planned to last until end of 2022. At each site, study will last until 26 months after the last randomization in that site.

Study procedures:

The treatment should be given at the time of randomization; participants will be followed for the duration of treatment (i.e. 2-4 months), and for 2 years after treatments is finished.

Follow up during treatment consists of 3 clinic visits for participants in all arms. At each visit, a pill count and monitoring of possible side effects will be performed.

Follow-up after treatment will consist of contacting participants by phone every 3 months for 2 years, to check for symptoms of active TB.

Outcomes definitions:

Primary outcomes:

1. Treatment completion (i.e. comparing how many people in each group completed treatment). Treatment completion is defined as taking at least 80% of the doses in 120% of the allowed time. The number of pills taken will be known by counting the pills dispensed and brought back by participants at each visit while they are on treatment.
2. Safety: Grade 3-5 adverse events that result in permanent discontinuation of study drug and are considered probably or possibly related to the study drug by an independent 3-member adjudication panel blinded to study treatment.

Secondary outcomes:

1. Safety: grade 1-2 adverse events that result in permanent discontinuation of study drug and are considered probably or possibly related to the study drug by the same independent 3-member adjudication panel.
2. Efficacy: comparing rates of active TB in the 26 months post-randomization

Statistical analyses:

There are two planned primary analyses, comparing each of the two intervention arms to the conventional arm: 1) Superiority of treatment completion, using a logistic regression; 2) Non-inferiority of safety, using a Poisson regression to compare the occurrence of the grade 3-5 adverse events. We will use the confidence interval approach, and compare the upper limit of the difference using a margin of 4%.

Given that some exclusion post randomization could occur (for example if drug sensitivity test (DST) results for the index case were not available at the time of randomization but later showed resistance to rifampin- their contacts would not be eligible for the study and would be subsequently be excluded), a modified intention to treat analysis will be used - with these valid post-randomization exclusions. A secondary analysis will be done among patients who completed therapy per protocol.

Other planned secondary analyses are: 1) Non-inferiority of completion. The maximum allowable difference will be 5%, with one-sided significance level; 2) Non-inferiority of grade 1-2 adverse events (in the same way as grade 3-5 adverse events done for primary analysis); 3) Comparison of incidence of active TB per 100 person-years of follow-up, in the 26 months post-randomization. All analyses will include adjustment for clustering by household. In stratified analysis, results will be presented by indication for LTBI treatment. Sensitivity analyses will be conducted where by analysis are stratified by study centre and by country.

Interim Analyses:

There will be at least two interim analyses of study regimen completion and of Grade 3-5 adverse events. The first analysis will be conducted after the first 150 participants have completed therapy, the second after 450 participants have completed therapy or sooner if there are concerns about excess toxicity with either high-dose arm. The Data and Safety Monitoring Board (DSMB) will be responsible to review the two planned interim analyses, as well as any unexpected Grade 4 adverse events, or deaths that could be related to study regimens. Rather than having a formal stopping rule, the decision to stop enrollment, would be made by the DSMB, based on the safety reports received and the results of interim analyses.

ELIGIBILITY:
Inclusion Criteria:

* Adults, and children aged 10 and older who weigh at least 25kg.
* Evidence of latent TB infection: positive tuberculin skin test (5mm or greater or 10mm or greater, based on National guidelines) or positive interferon gamma release assay.
* Eligible to take latent TB treatment according to Canadian guidelines in the Canadian sites, and according to World Health Organization (WHO) guidelines in the international sites (this includes household contacts, other contacts, HIV infected, other causes of immune suppression, fibronodular disease on chest-x ray (CXR), or other indication).

Exclusion Criteria:

* Children aged 0-9 and children aged 10 or older who weigh less than 25kg
* Pregnancy
* Baseline AST or ALT that is at least 3 times higher than upper limit of normal
* Baseline Grade 3-4 abnormalities of hematological tests (WBC, platelets or hemoglobin).
* Prior treatment for latent or active TB.
* Rifampin contra-indicated - due to potential drug interactions that are considered too important, or difficult to manage, by health care provider; or due to history of allergy/ hypersensitivity to rifampin, rifabutin or rifapentine.
* Household contacts of index TB patients with confirmed, or suspected rifampin resistant TB.

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1368 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment completion (taking 80% of doses within 120% of allowed time) | 2 months from randomization for participants in the two intervention arms and 4 months for the control arm.
  Completion will be defined as taking 80% of doses within 120% of allowed time (48 doses within 72 days for the two-month regimens, and 96 doses within 144 days for the 4-month regimen).
Safety measured by Grade 3 to 5 adverse events | 2 months plus 2 weeks in the intervention arms; 4 months plus 2 weeks in the control arm.
  Grade 3 to 5 adverse events (and Grade 1-2 rash) which result in permanent discontinuation of the study drug, and that are considered probably or possibly related to the study drug by the majority of a three-member independent and blinded Adverse Events panel.

SECONDARY OUTCOMES:
Safety measured by Grade 1 to 2 adverse events | 2 months plus 2 weeks in the intervention arms; 4 months plus 2 weeks in the control arm.
  Grade 1 to 2 adverse events which result in permanent discontinuation of the study drug and are considered probably or possibly related to the study drug by the adverse events panel.
Efficacy measured during follow-up visits and telephone calls | 26 months from randomization in all arms.
  Active TB - symptoms will be ascertained monthly by direct questioning during treatment phase follow-up visits, and by telephone call every 3 months up to 26 months after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Dick Menzies, Principal Investigator — RI-MUHC
Locations (9):
- Canada (4):
  - Unviversity of Calgary, Calgary, Alberta
  - The Governors of the University of Alberta, Edmonton, Alberta
  - BCCDC TB clinic, Vancouver, British Columbia
  - MUHC, Montreal, Quebec
- Universitas Padjadjaran, Klinik Penelitian Tuberculosis (TB research clinic), Bandung, Indonesia
- Vietnam (4):
  - Hai Ba Trung District Health Center, No. 16B, Hà Nội
  - Hanoi Lung Hospital, Hà Nội
  - Nam Tu Liem District Health Center, No. 3, Hà Nội
  - Phoi Viet TB and Respiratory Diseases Clinic., Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Protocol and consent form will be available for data sharing once approved by research ethical review board. A detailed plan for data sharing of other study documents and/or data is under definition and will be posted during the trial.
Supporting Information: Study Protocol, ICF
Time Frame: Protocol and consent form will be available once approval is received from the research ethical board and will remain available.
Access Criteria: Access criteria will be specified in the plan for data sharing, once available.

REFERENCES:
- [Background] Aarnoutse RE, Kibiki GS, Reither K, Semvua HH, Haraka F, Mtabho CM, Mpagama SG, van den Boogaard J, Sumari-de Boer IM, Magis-Escurra C, Wattenberg M, Logger JGM, Te Brake LHM, Hoelscher M, Gillespie SH, Colbers A, Phillips PPJ, Plemper van Balen G, Boeree MJ; PanACEA Consortium. Pharmacokinetics, Tolerability, and Bacteriological Response of Rifampin Administered at 600, 900, and 1,200 Milligrams Daily in Patients with Pulmonary Tuberculosis. Antimicrob Agents Chemother. 2017 Oct 24;61(11):e01054-17. doi: 10.1128/AAC.01054-17. Print 2017 Nov. PMID 28827417
- [Background] Boeree MJ, Heinrich N, Aarnoutse R, Diacon AH, Dawson R, Rehal S, Kibiki GS, Churchyard G, Sanne I, Ntinginya NE, Minja LT, Hunt RD, Charalambous S, Hanekom M, Semvua HH, Mpagama SG, Manyama C, Mtafya B, Reither K, Wallis RS, Venter A, Narunsky K, Mekota A, Henne S, Colbers A, van Balen GP, Gillespie SH, Phillips PPJ, Hoelscher M; PanACEA consortium. High-dose rifampicin, moxifloxacin, and SQ109 for treating tuberculosis: a multi-arm, multi-stage randomised controlled trial. Lancet Infect Dis. 2017 Jan;17(1):39-49. doi: 10.1016/S1473-3099(16)30274-2. Epub 2016 Oct 26. PMID 28100438
- [Background] Dian S, Yunivita V, Ganiem AR, Pramaesya T, Chaidir L, Wahyudi K, Achmad TH, Colbers A, Te Brake L, van Crevel R, Ruslami R, Aarnoutse R. Double-Blind, Randomized, Placebo-Controlled Phase II Dose-Finding Study To Evaluate High-Dose Rifampin for Tuberculous Meningitis. Antimicrob Agents Chemother. 2018 Nov 26;62(12):e01014-18. doi: 10.1128/AAC.01014-18. Print 2018 Dec. PMID 30224533
- [Background] Jindani A, Borgulya G, de Patino IW, Gonzales T, de Fernandes RA, Shrestha B, Atwine D, Bonnet M, Burgos M, Dubash F, Patel N, Checkley AM, Harrison TS, Mitchison D; International Consortium for Trials of Chemotherapeutic Agents in Tuberculosis, St George's University of London. A randomised Phase II trial to evaluate the toxicity of high-dose rifampicin to treat pulmonary tuberculosis. Int J Tuberc Lung Dis. 2016 Jun;20(6):832-8. doi: 10.5588/ijtld.15.0577. PMID 27155189
- [Background] Ruslami R, Ganiem AR, Dian S, Apriani L, Achmad TH, van der Ven AJ, Borm G, Aarnoutse RE, van Crevel R. Intensified regimen containing rifampicin and moxifloxacin for tuberculous meningitis: an open-label, randomised controlled phase 2 trial. Lancet Infect Dis. 2013 Jan;13(1):27-35. doi: 10.1016/S1473-3099(12)70264-5. Epub 2012 Oct 25. PMID 23103177
- [Background] Ruslami R, Nijland HM, Alisjahbana B, Parwati I, van Crevel R, Aarnoutse RE. Pharmacokinetics and tolerability of a higher rifampin dose versus the standard dose in pulmonary tuberculosis patients. Antimicrob Agents Chemother. 2007 Jul;51(7):2546-51. doi: 10.1128/AAC.01550-06. Epub 2007 Apr 23. PMID 17452486
- [Background] Swindells S, Ramchandani R, Gupta A, Benson CA, Leon-Cruz J, Mwelase N, Jean Juste MA, Lama JR, Valencia J, Omoz-Oarhe A, Supparatpinyo K, Masheto G, Mohapi L, da Silva Escada RO, Mawlana S, Banda P, Severe P, Hakim J, Kanyama C, Langat D, Moran L, Andersen J, Fletcher CV, Nuermberger E, Chaisson RE; BRIEF TB/A5279 Study Team. One Month of Rifapentine plus Isoniazid to Prevent HIV-Related Tuberculosis. N Engl J Med. 2019 Mar 14;380(11):1001-1011. doi: 10.1056/NEJMoa1806808. PMID 30865794
- [Background] Velasquez GE, Brooks MB, Coit JM, Pertinez H, Vargas Vasquez D, Sanchez Garavito E, Calderon RI, Jimenez J, Tintaya K, Peloquin CA, Osso E, Tierney DB, Seung KJ, Lecca L, Davies GR, Mitnick CD. Efficacy and Safety of High-Dose Rifampin in Pulmonary Tuberculosis. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2018 Sep 1;198(5):657-666. doi: 10.1164/rccm.201712-2524OC. PMID 29954183
- [Background] Yunivita V, Dian S, Ganiem AR, Hayati E, Hanggono Achmad T, Purnama Dewi A, Teulen M, Meijerhof-Jager P, van Crevel R, Aarnoutse R, Ruslami R. Pharmacokinetics and safety/tolerability of higher oral and intravenous doses of rifampicin in adult tuberculous meningitis patients. Int J Antimicrob Agents. 2016 Oct;48(4):415-21. doi: 10.1016/j.ijantimicag.2016.06.016. Epub 2016 Jul 26. PMID 27526979
- [Derived] Ruslami R, Fregonese F, Apriani L, Barss L, Bedingfield N, Chiang V, Cook VJ, Fisher D, Flores E, Fox GJ, Johnston J, Lim RK, Long R, Paulsen C, Nguyen TA, Nhung NV, Gibson D, Valiquette C, Benedetti A, Menzies D. High-dose, short-duration versus standard rifampicin for tuberculosis preventive treatment: a partially blinded, three-arm, non-inferiority, randomised, controlled trial. Lancet Respir Med. 2024 Jun;12(6):433-443. doi: 10.1016/S2213-2600(24)00076-6. Epub 2024 Mar 26. PMID 38552659
- [Derived] Fregonese F, Apriani L, Barss L, Benedetti A, Cook V, Fisher D, Fox GJ, Johnston J, Long R, Nguyen TA, Nguyen VN, Ruslami R, Menzies D. High dose rifampin for 2 months vs standard dose rifampin for 4 months, to treat TB infection: Protocol of a 3-arm randomized trial (2R2). PLoS One. 2023 Feb 2;18(2):e0278087. doi: 10.1371/journal.pone.0278087. eCollection 2023. PMID 36730240